CLINICAL TRIAL: NCT04957979
Title: Comparing Two Approaches to Care Coordination for High-Cost/High-Need Patients in Primary Care
Brief Title: Minnesota Care Coordination Effectiveness Study
Acronym: MNCARES
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Minnesota Department of Health (Other Government); MN Community Measurement (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19-110; IHS-2019C1-15625 (Other: Patient Centered Outcomes Research Institute)
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Chronic Disease; Multi-morbidity; Care Coordination
Keywords: Care Coordination; Quality of Care; Health Care Utilization
MeSH Terms: conditions — Chronic Disease; Patient Acceptance of Health Care | interventions — Nursing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nursing/Medical Model of Care Coordination: Someone with medical/nursing training coordinates involvement of various medical resources and provides patients with education, self-management support, and referrals to community resources.
  Interventions: Other: Nursing/Medical Model of Care Coordination
- Medical/Social Model of Care Coordination: In addition to the services provided in the Medical/Nursing Model, a social worker by education has dedicated FTE as a member of the care team at the clinic, providing some direct services for care coordination patients and either spending some time on-site or in regular communication with its clinicians in addition to providing social work services.
  Interventions: Other: Medical/Social Model of Care Coordination

INTERVENTIONS:
Other: Nursing/Medical Model of Care Coordination — No social worker on the clinic's care coordination team.
  Services provided:
  * Coordinated medical care for patients
  * Patient education
  * Assistance in developing care plan
  * Support for patient self-management
  * Referrals for continuing care
  * Referral to community resources
  * Referral to mental health services if needed or requested
  * Referral to interventional counseling for behavioral health issues
  Groups: Nursing/Medical Model of Care Coordination
Other: Medical/Social Model of Care Coordination — Social worker is part of the clinic's care coordination team.
  * Need not be licensed as a social worker
  * Must have time dedicated to care coordination for a specific clinic or clinics
  * Must interact with individual patients to provide them with services
  * Must interact with individual clinicians about their individual patients in care coordination
  Services provided:
  * Coordinated medical care for patients
  * Patient education
  * Assistance in developing care plan
  * Support for patient self-management
  * Assistance with referrals for continuing care
  * Assessment and plan to address social and resource needs including housing, transportation or financial needs; Assist patient in locating and obtaining needed community resources
  * Assistance with identifying and addressing psychological/emotional issues and referrals as needed
  * Interventional counseling for behavioral health issues or referrals to interventional counseling, depending on licensure
  Groups: Medical/Social Model of Care Coordination

SUMMARY:
Medical care has improved greatly over the past 50 years. Treatments for most medical conditions can help us lead longer and healthier lives, but there are still problems. Many patients with two or more conditions see many different doctors and sometimes take more medications than needed. These patients can feel lost and confused. In addition, non-medical issues involving housing, food, transportation, employment, income, support from others, and language barriers can have a large impact on our health.

In Minnesota, many primary care clinics are using a method called care coordination to improve the health of patients who have a number of chronic diseases (some examples of chronic diseases include diabetes, heart disease, asthma and depression). With care coordination, a nurse in the clinic helps the various doctors, clinics, and specialists to work together, in the interest of the patient. In some clinics, a social worker also helps with care coordination. These social workers help with issues like housing, transportation, or employment. Care coordination can help reduce patient confusion. It also can improve health and lower patient burdens and costs of getting medical care.

To help find out what types of care coordination are most successful, we are proposing a study. Our plan is to track the health of patients receiving care coordination and compare two types:

A. Care coordination done by a nurse or other clinic staff B. Care coordination where a licensed social worker also assists the patient

In this study, we will measure many things, including:

1. Control of chronic conditions like diabetes, heart disease, asthma, and depression
2. Hospitalizations
3. Emergency department visits
4. Use of medications and diagnostic tests
5. Use of specialty care
6. General health status
7. Patient satisfaction and access to care
8. Use of shared decision-making (where the doctor and the patient make treatment decisions together)
9. Patient burden (how much time and effort the patient spends trying to get healthy)
10. Patients' out-of-pocket medical costs

This project will be important to patients because it could reduce confusion and fragmented care while improving all the items above. Those improvements will be more likely because this project takes advantage of engagement with patients and others. We have four patient partners who will help conduct the study and interpret and broadly share the results. The project was developed with the input from patients, clinic leaders, people from state government, and experts on health and quality care.

By measuring a wide variety of outcomes for the adults receiving coordination services in these clinics, we hope to identify the specific actionable information that will allow these and other clinics to improve their services for these patients with complex needs.

Throughout the project, we will communicate our findings to clinics and health systems. As a result, many people may receive better care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Historical Cohort: Receiving care coordination services in a participating clinic with a care coordination start date between January 2018 and February 2019
* Primary Cohort: Receiving care coordination services in a participating clinic with a care coordination start date between January 2021 and December 2021
* Currently insured by the MN Department of Human Services (DHS), Blue Cross Blue Shield MN (BCBS), UCare, or HealthPartners (HP) (for utilization outcomes only)
* Consents to participate in interview or responds to a survey (for those data collection events only)

Exclusion Criteria:

* Cannot complete an interview in English (interviews only)
* Cannot complete a survey in English, Spanish, Somali, or Hmong (for interviews only, reflecting most prevalent languages in MN)
* On a known research exclusion list

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants are patients receiving care coordination in Minnesota's Health Care Homes certified adult primary care clinics, starting during the specified date ranges.
Sampling Method: Non-Probability Sample
Enrollment: 25507 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leif I Solberg, MD, Principal Investigator — HealthPartners Institute; Steven P Dehmer, PhD, Principal Investigator — HealthPartners Institute
Locations (3):
- United States (3):
  - MN Community Measurement, Minneapolis, Minnesota
  - HealthPartners Institute, Minneapolis, Minnesota
  - Minnesota Department of Health (MDH), Saint Paul, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinic recruitment was performed in late 2020. Participating clinics identified patients for trial inclusion between 2021 and 2023. Patient surveys were administered in late 2022 (Historical Cohort) and late 2023 (Primary Cohort).
Pre-assignment Details: This is an observational trial so patients were identified for inclusion in the trial by their home clinics. Each home clinic was classified to one of the two comparison arms based on the care models they were already performing, and all patients receiving care in that clinic were assigned to that arm. No patients identified by clinics that met inclusion criteria were excluded.
Units Other Than Participants: Clinics
Groups:
- Historical Cohort: Medical/Nursing Model: Patients starting care coordination in participating clinics between January 2018 and February 2019.
  Someone with medical/nursing training coordinates involvement of various medical resources and provides patients with education, self-management support, and referrals to community resources.
  Nursing/Medical Model of Care Coordination: No social worker on the clinic's care coordination team.
  Services provided:
  * Coordinated medical care for patients
  * Patient education
  * Assistance in developing care plan
  * Support for patient self-management
  * Referrals for continuing care
  * Referral to community resources
  * Referral to mental health services if needed or requested
  * Referral to interventional counseling for behavioral health issues
- Historical Cohort: Medical/Social Model: Patients starting care coordination in participating clinics between January 2018 and February 2019.
  In addition to the services provided in the Medical/Nursing Model, a social worker by education has dedicated FTE as a member of the care team at the clinic, providing some direct services for care coordination patients and either spending some time on-site or in regular communication with its clinicians in addition to providing social work services.
  Medical/Social Model of Care Coordination: Social worker is part of the clinic's care coordination team.
  * Need not be licensed as a social worker
  * Must have time dedicated to care coordination for a specific clinic or clinics
  * Must interact with individual patients to provide them with services
  * Must interact with individual clinicians about their individual patients in care coordination
  Services provided:
  * Coordinated medical care for patients
  * Patient education
  * Assistance in developing care plan
  * Support for patient self-management
  * Assistance with referrals for continuing care
  * Assessment and plan to address social and resource needs including housing, transportation or financial needs; Assist patient in locating and obtaining needed community resources
  * Assistance with identifying and addressing psychological/emotional issues and referrals as needed
  * Interventional counseling for behavioral health issues or referrals to interventional counseling, depending on licensure
- Primary Cohort: Medical/Nursing Model: Patients starting care coordination in participating clinics between January and December 2021.
  Someone with medical/nursing training coordinates involvement of various medical resources and provides patients with education, self-management support, and referrals to community resources.
  Nursing/Medical Model of Care Coordination: No social worker on the clinic's care coordination team.
  Services provided:
  * Coordinated medical care for patients
  * Patient education
  * Assistance in developing care plan
  * Support for patient self-management
  * Referrals for continuing care
  * Referral to community resources
  * Referral to mental health services if needed or requested
  * Referral to interventional counseling for behavioral health issues
- Primary Cohort: Medical/Social Model: Patients starting care coordination in participating clinics between January-December 2021.
  In addition to the services provided in the Medical/Nursing Model, a social worker by education has dedicated FTE as a member of the care team at the clinic, providing some direct services for care coordination patients and either spending some time on-site or in regular communication with its clinicians in addition to providing social work services.
  Medical/Social Model of Care Coordination: Social worker is part of the clinic's care coordination team.
  * Need not be licensed as a social worker
  * Must have time dedicated to care coordination for a specific clinic or clinics
  * Must interact with individual patients to provide them with services
  * Must interact with individual clinicians about their individual patients in care coordination
  Services provided:
  * Coordinated medical care for patients
  * Patient education
  * Assistance in developing care plan
  * Support for patient self-management
  * Assistance with referrals for continuing care
  * Assessment and plan to address social and resource needs including housing, transportation or financial needs; Assist patient in locating and obtaining needed community resources
  * Assistance with identifying and addressing psychological/emotional issues and referrals as needed
  * Interventional counseling for behavioral health issues or referrals to interventional counseling, depending on licensure
Period: Overall Study
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Started | 4110; 107 Clinics | 8721; 122 Clinics | 3572; 151 Clinics | 9104; 129 Clinics
Completed | 4110; 107 Clinics | 8721; 122 Clinics | 3572; 151 Clinics | 9104; 129 Clinics
Not Completed | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics | 0; 0 Clinics

BASELINE CHARACTERISTICS:
Population: Baseline population is the population of patients identified by care systems meeting study eligibility criteria.
Groups:
- Primary Cohort: Medical/Nursing Model: Patients starting care coordination in participating clinics between January-December 2021.
  Someone with medical/nursing training coordinates involvement of various medical resources and provides patients with education, self-management support, and referrals to community resources.
  Nursing/Medical Model of Care Coordination: No social worker on the clinic's care coordination team.
  Services provided:
  * Coordinated medical care for patients
  * Patient education
  * Assistance in developing care plan
  * Support for patient self-management
  * Referrals for continuing care
  * Referral to community resources
  * Referral to mental health services if needed or requested
  * Referral to interventional counseling for behavioral health issues
- Total: Total of all reporting groups
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model | Total
Number analyzed (Participants) | 4110 | 8721 | 3572 | 9104 | 25507
Age, Continuous [Mean (Standard Deviation); unit: years] — As documented in the EHR, at start of care coordination
  years | 63 (18) | 62 (19) | 62 (18) | 63 (18) | 62 (19)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2456 | 5418 | 2250 | 5659 | 15783
  Male | 1654 | 3299 | 1308 | 3445 | 9706
  Unknown | 0 | 4 | 14 | 0 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — As documented in the EHR
  Participants
    Hispanic or Latino | 107 | 271 | 202 | 285 | 865
    Not Hispanic or Latino | 3540 | 7980 | 2642 | 7791 | 21953
    Unknown or Not Reported | 463 | 470 | 728 | 1028 | 2689
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — As documented in the EHR
  Participants
    American Indian or Alaska Native | 34 | 214 | 76 | 272 | 596
    Asian | 112 | 1090 | 681 | 1486 | 3369
    Black or African American | 196 | 944 | 198 | 1185 | 2523
    Hispanic or Latino | 56 | 149 | 102 | 24 | 331
    Native Hawaiian/Other Pacific Islander | 1 | 10 | 11 | 17 | 39
    Other | 23 | 87 | 57 | 46 | 213
    White | 3625 | 5924 | 2335 | 5776 | 17660
    Unknown or Choose not to answer | 63 | 303 | 112 | 298 | 776
Primary Language [Count of Participants; unit: Participants] — As indicated in the EHR for patients requesting language interpreter services
  Participants
    English | 3905 | 7071 | 3211 | 7244 | 21431
    Hmong | 11 | 263 | 15 | 349 | 638
    Somali | 26 | 224 | 39 | 226 | 515
    Spanish | 62 | 176 | 158 | 185 | 581
    Other | 90 | 953 | 115 | 1092 | 2250
    Unknown or Choose not to answer | 16 | 34 | 34 | 8 | 92
Country of Origin [Count of Participants; unit: Participants] — As documented in the EHR
  Participants
    United States | 3019 | 5780 | 2552 | 6133 | 17484
    Non-US country | 198 | 1787 | 217 | 2062 | 4264
    Unknown or Choose not to answer | 893 | 1154 | 803 | 909 | 3759
Insurance coverage [Count of Participants; unit: Participants] — As documented in EHR
  Participants
    Government-sponsored insurance plans | 800 | 3950 | 1076 | 4519 | 10345
    Non-government sponsored insurance plans | 3310 | 4771 | 2496 | 4585 | 15162
Number of chronic conditions [Count of Participants; unit: Participants] — As documented in EHR problem list
  Participants
    0 | 322 | 285 | 295 | 346 | 1248
    1 | 233 | 369 | 186 | 420 | 1208
    2 | 267 | 595 | 257 | 522 | 1641
    3-4 | 711 | 1496 | 601 | 1371 | 4179
    5-6 | 908 | 1571 | 708 | 1596 | 4783
    7-8 | 741 | 1490 | 641 | 1623 | 4495
    9-10 | 466 | 1182 | 423 | 1286 | 3357
    11+ | 462 | 1733 | 461 | 1940 | 4596
Prevalent chronic conditions [Count of Participants; unit: Participants] — As documented in the EHR problem list, with at least 20% prevalence in a study subgroup
  Participants
    Anemia | 696 | 2114 | 629 | 2360 | 5799
    Anxiety disorders | 1403 | 3833 | 1350 | 3968 | 10554
    Blindness and vision loss | 1088 | 2723 | 941 | 3169 | 7921
    Chronic kidney disease | 962 | 2556 | 817 | 2912 | 7247
    Depressive disorders | 1481 | 4026 | 1341 | 4298 | 11146
    Diabetes | 2005 | 4129 | 1764 | 4379 | 12277
    Drug use disorders | 613 | 2004 | 653 | 2112 | 5382
    Hyperlipidemia | 2282 | 4881 | 1872 | 5097 | 14132
    Hypertension | 2412 | 5308 | 1992 | 5529 | 15241
    Ischaemic heart disease | 766 | 1909 | 678 | 1949 | 5302
    Low back pain | 1040 | 2811 | 968 | 3172 | 7991
    Osteoarthritis | 1182 | 2832 | 1076 | 3166 | 8256

OUTCOME MEASURES:

1. Primary Outcome: Change in Composite Measure of Care Quality
Description: The analytic outcome is defined as the absolute change in the percentage of eligible care quality measures met by a patient in the year before and after care coordination initiation. The composite measure of care quality is calculated as the percentage of all applicable care quality measures a patient meets based on clinical guidelines, including control of blood pressure, cardiovascular disease, diabetes, asthma, depression, and cancer screening. Criteria for each of the components was assessed using health outcomes from EHR and insurance claims to capture occurrence and timing of recommended screenings. A positive change (post % - pre % > 0) reflects an improvement in the percentage of care quality measures met, while a negative change indicates a decline.
Time Frame: 12 months pre- and post- initiation of care coordination
Population: Patients included in analytic comparison if they qualify for at least one care quality outcome in both the year pre- and post-care coordination initiation.
Measure: Mean (Standard Deviation); unit: Change in percent
Groups:
- Primary Cohort: Medical/Nursing Model: Patients starting care coordination in participating clinics between January 2021 and December 2021.
  Someone with medical/nursing training coordinates involvement of various medical resources and provides patients with education, self-management support, and referrals to community resources.
  Nursing/Medical Model of Care Coordination: No social worker on the clinic's care coordination team.
  Services provided:
  * Coordinated medical care for patients
  * Patient education
  * Assistance in developing care plan
  * Support for patient self-management
  * Referrals for continuing care
  * Referral to community resources
  * Referral to mental health services if needed or requested
  * Referral to interventional counseling for behavioral health issues
- Primary Cohort: Medical/Social Model: Patients starting care coordination in participating clinics between January 2021 and December 2021.
  In addition to the services provided in the Medical/Nursing Model, a social worker by education has dedicated FTE as a member of the care team at the clinic, providing some direct services for care coordination patients and either spending some time on-site or in regular communication with its clinicians in addition to providing social work services.
  Medical/Social Model of Care Coordination: Social worker is part of the clinic's care coordination team.
  * Need not be licensed as a social worker
  * Must have time dedicated to care coordination for a specific clinic or clinics
  * Must interact with individual patients to provide them with services
  * Must interact with individual clinicians about their individual patients in care coordination
  Services provided:
  * Coordinated medical care for patients
  * Patient education
  * Assistance in developing care plan
  * Support for patient self-management
  * Assistance with referrals for continuing care
  * Assessment and plan to address social and resource needs including housing, transportation or financial needs; Assist patient in locating and obtaining needed community resources
  * Assistance with identifying and addressing psychological/emotional issues and referrals as needed
  * Interventional counseling for behavioral health issues or referrals to interventional counseling, depending on licensure
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 2514 | 5326 | 2097 | 5546
Change in percent | 7.0 (31.2) | 4.5 (34.3) | 5.9 (31.1) | 5.9 (35.7)
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Null hypothesis: Average change in composite care quality outcome is not different between patients receiving care in Medical/Nursing Model clinics and those receiving care in Medical/Social Model clinics; Test type: Superiority; p = 0.19, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Adjusted for patient demographics, comorbidities, clinic characteristics, and includes random effect for clustering within clinic; Mean Difference (Net) = -1.6, 95% CI 2-sided [-4.1 to 0.1] — Negative value represents smaller change in Medical/Social clinics as compared to Medical/Nursing
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.005, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -3.3, 95% CI 2-sided [-5.6 to -1.0] — Negative value represents smaller change in Medical/Social clinics as compared to Medical/Nursing

2. Primary Outcome: Change in Annual Number of Emergency Department Visits
Description: Change in # of encounters with CPT-4 E&M codes (99281-99288) at emergency departments across the year before and year after care coordination initiation per 100 people. Negative values of change represent improvement, positive values represent a increase in number of admissions.
Time Frame: 12 months pre and post start of care coordination
Population: Patients included in analytic comparison if they were covered by participating insurers in both the year pre- and post-care coordination initiation.
Measure: Mean (Standard Deviation); unit: Change in encounters per 100 people per
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 767 | 2487 | 925 | 3811
Change in encounters per 100 people per | -0.261 (127.8) | -0.523 (174.5) | -5.51 (185.3) | -2.97 (248.8)
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Generalized Linear Mixed Models with Poisson link function. Pre-care coordination measures were included as an independent variable when modeling post-measures to capture change related to care coordination initiation; Test type: Superiority; p = 0.02, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 1, analysis 1]; Incidence Rate Ratio = 1.28, 95% CI 2-sided [1.04 to 1.58] — Values > 1.0 represents higher rates post-care coordination in Medical/Social clinics as compared to Medical/Nursing
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.45, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 1, analysis 1]; Incidence Rate Ratio = 1.09, 95% CI 2-sided [0.868 to 1.38] — Values > 1.0 represents higher rates post-care coordination in Medical/Social clinics as compared to Medical/Nursing

3. Primary Outcome: Change in Annual Number of Inpatient Hospitalizations
Description: Change in # of hospital inpatient admissions ≥ 1 days across the year before and year after care coordination initiation per 100 people. Negative values of change represent improvement, positive values represent a increase in number of admissions.
Time Frame: 12 months pre and post start of care coordination
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in encounters per 100 people per
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 767 | 2487 | 925 | 3811
Change in encounters per 100 people per | -1.173 (106.6) | 7.197 (178.4) | -7.459 (164.2) | -4.828 (161.3)
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.01, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 1, analysis 1]; Incidence Rate Ratio = 1.35, 95% CI 2-sided [1.08 to 1.69] — Values > 1.0 represents higher rates post-care coordination in Medical/Social clinics as compared to Medical/Nursing
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.08, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 1, analysis 1]; Incidence Rate Ratio = 1.33, 95% CI 2-sided [0.969 to 1.81] — Values > 1.0 represents higher rates post-care coordination in Medical/Social clinics as compared to Medical/Nursing

4. Primary Outcome: General Health Status - Top Box Scoring
Description: Percentage of patients reporting Excellent, Very Good, or Good when asked to rate general health status on 5-level Likert Scale (NHIS)
Time Frame: 6 to 18 months after start of care coordination
Population: Patients included in analytic comparison if they responded to patient survey sent at least 6 months after care coordination initiation date and provided answer to relevant survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 335 | 486 | 929 | 1841
Participants | 221 | 365 | 609 | 1002
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Generalized Linear Mixed Models with Binomial link function; Test type: Superiority; p = 0.0001, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.51 to 0.81] — Values > 1.0 represents higher likelihood of positive rating in Medical/Social clinics as compared to Medical/Nursing
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Generalized Linear Mixed Models with Binomial link function; Test type: Superiority; p = 0.32, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.84 to 1.72] — Values > 1.0 represents higher likelihood of positive rating in Medical/Social clinics as compared to Medical/Nursing

5. Primary Outcome: Rating of Primary Care Clinic - Top Box
Description: Percentage of patients reporting 9 or 10 when asked to rate primary care clinic (CG-CAHPS)
Time Frame: 6 to 18 months after start of care coordination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 329 | 469 | 914 | 1825
Participants | 188 | 235 | 480 | 898
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Generalized Linear Mixed Models with Binomial link function; Test type: Superiority; p = 0.14, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.69 to 1.05] — Values > 1.0 represents higher likelihood of positive rating in Medical/Social clinics as compared to Medical/Nursing
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Generalized Linear Mixed Models with Binomial link function; Test type: Superiority; p = 0.12, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.51 to 1.08] — Values > 1.0 represents higher likelihood of positive rating in Medical/Social clinics as compared to Medical/Nursing

6. Secondary Outcome: Change in Percent of Patients Meeting Asthma Care at Goal
Description: The analytic outcome is defined as the absolute change in the percentage of eligible patients (those with a current asthma diagnosis) demonstrating asthma control (Asthma Control Test (ACT) score <19) within each arm in the year before and after care coordination initiation. A positive change reflects an improvement in the percentage of eligible patients with asthma control while a negative change indicates a decline.
Time Frame: 12 months pre and post start of care coordination
Population: Patients included in analytic comparison if they have a diagnosis of asthma in both the year pre- and post-care coordination initiation.
Measure: Number; unit: Change in percent
Groups:
- Historical Cohort - Nursing/Medical Model of Care Coordination: Patients starting care coordination in participating clinics between January 2018 and February 2019.
  Someone with medical/nursing training coordinates involvement of various medical resources and provides patients with education, self-management support, and referrals to community resources.
  Nursing/Medical Model of Care Coordination: No social worker on the clinic's care coordination team.
  Services provided:
  * Coordinated medical care for patients
  * Patient education
  * Assistance in developing care plan
  * Support for patient self-management
  * Referrals for continuing care
  * Referral to community resources
  * Referral to mental health services if needed or requested
  * Referral to interventional counseling for behavioral health issues
- Historical Cohort - Medical/Social Model of Care Coordination: Patients starting care coordination in participating clinics between January 2018 and February 2019.
  In addition to the services provided in the Medical/Nursing Model, a social worker by education has dedicated FTE as a member of the care team at the clinic, providing some direct services for care coordination patients and either spending some time on-site or in regular communication with its clinicians in addition to providing social work services.
  Medical/Social Model of Care Coordination: Social worker is part of the clinic's care coordination team.
  * Need not be licensed as a social worker
  * Must have time dedicated to care coordination for a specific clinic or clinics
  * Must interact with individual patients to provide them with services
  * Must interact with individual clinicians about their individual patients in care coordination
  Services provided:
  * Coordinated medical care for patients
  * Patient education
  * Assistance in developing care plan
  * Support for patient self-management
  * Assistance with referrals for continuing care
  * Assessment and plan to address social and resource needs including housing, transportation or financial needs; Assist patient in locating and obtaining needed community resources
  * Assistance with identifying and addressing psychological/emotional issues and referrals as needed
  * Interventional counseling for behavioral health issues or referrals to interventional counseling, depending on licensure
- Primary Cohort - Nursing/Medical Model of Care Coordination: Patients starting care coordination in participating clinics between January 2021 and December 2021.
  Someone with medical/nursing training coordinates involvement of various medical resources and provides patients with education, self-management support, and referrals to community resources.
  Nursing/Medical Model of Care Coordination: No social worker on the clinic's care coordination team.
  Services provided:
  * Coordinated medical care for patients
  * Patient education
  * Assistance in developing care plan
  * Support for patient self-management
  * Referrals for continuing care
  * Referral to community resources
  * Referral to mental health services if needed or requested
  * Referral to interventional counseling for behavioral health issues
- Primary Cohort - Medical/Social Model of Care Coordination: Patients starting care coordination in participating clinics between January 2021 and December 2021.
  In addition to the services provided in the Medical/Nursing Model, a social worker by education has dedicated FTE as a member of the care team at the clinic, providing some direct services for care coordination patients and either spending some time on-site or in regular communication with its clinicians in addition to providing social work services.
  Medical/Social Model of Care Coordination: Social worker is part of the clinic's care coordination team.
  * Need not be licensed as a social worker
  * Must have time dedicated to care coordination for a specific clinic or clinics
  * Must interact with individual patients to provide them with services
  * Must interact with individual clinicians about their individual patients in care coordination
  Services provided:
  * Coordinated medical care for patients
  * Patient education
  * Assistance in developing care plan
  * Support for patient self-management
  * Assistance with referrals for continuing care
  * Assessment and plan to address social and resource needs including housing, transportation or financial needs; Assist patient in locating and obtaining needed community resources
  * Assistance with identifying and addressing psychological/emotional issues and referrals as needed
  * Interventional counseling for behavioral health issues or referrals to interventional counseling, depending on licensure
Arm/Group | Historical Cohort - Nursing/Medical Model of Care Coordination | Historical Cohort - Medical/Social Model of Care Coordination | Primary Cohort - Nursing/Medical Model of Care Coordination | Primary Cohort - Medical/Social Model of Care Coordination
Number analyzed (Participants) | 43 | 117 | 28 | 136
Change in percent | -2.3 | -2.6 | -7.1 | -6.6
Statistical Analysis 1: Comparison: Primary Cohort - Nursing/Medical Model of Care Coordination vs Primary Cohort - Medical/Social Model of Care Coordination; Test type: Superiority; p = 0.914, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Binomial link function. Estimation parameter is the interaction between Time (post vs pre) and Care Model (Medical/Social vs Medical Nursing); Odds Ratio (OR) = 1.086, 95% CI 2-sided [0.243 to 4.861] — Values > 1.0 represents larger improvement pre to post-care coordination in likelihood of specific care quality outcome for patients in Medical/Social clinics as compared to those in Medical/Nursing
Statistical Analysis 2: Comparison: Historical Cohort - Nursing/Medical Model of Care Coordination vs Historical Cohort - Medical/Social Model of Care Coordination; Test type: Superiority; p = 0.987, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 1.009, 95% CI 2-sided [0.327 to 3.114] — [estimate comment as in outcome 6, analysis 1]

7. Secondary Outcome: Change in Percent of Patients Meeting Breast Cancer Screening Criteria
Description: Screening criteria defined as mammogram within the last 2 years.
Time Frame: 12 months pre and post start of care coordination
Population: Patients included in analytic comparison if they were women, 50-74 years old, and covered by participating insurer in both the year pre- and post-care coordination initiation
Measure: Number; unit: percentage of patients
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 396 | 1351 | 410 | 1420
percentage of patients | 2.8 | -0.4 | 0.2 | 4.7
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p = 0.204, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 1.257, 95% CI 2-sided [0.883 to 1.79] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.04, Mixed Models Analysis; Odds Ratio (OR) = 0.399, 95% CI 2-sided [0.166 to 0.958]

8. Secondary Outcome: Change in Percent of Patients Meeting Colorectal Cancer Screening (Up-to-date)
Description: Screening criteria defined as approved screening test within the last 1 to 10 years depending on type of test and current recomendations.
Time Frame: 12 months pre and post start of care coordination
Population: Patients included in analytic comparison if they were 50-75 years old and had available claims data the year pre- and post-care coordination initiation.
Measure: Number; unit: percentage of patients
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 2146 | 4428 | 1790 | 4442
percentage of patients | 3.3 | 2.0 | 3.2 | 4.2
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p = 0.302, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 1.257, 95% CI 2-sided [0.814 to 1.939] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.192, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.647 to 1.092] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: Change in Percent of Patients Meeting Chlamydia Screening (Up-to-date)
Description: Screening criteria defined as a screening test for chlamydia within the last year.
Time Frame: 12 months pre and post start of care coordination
Population: Patients included in analytic comparison if they were women and 16-24 years old and covered by participating insurer the year pre- and post-care coordination initiation.
Measure: Number; unit: percentage of patients
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 40 | 47 | 17 | 54
percentage of patients | -7.5 | 2.1 | 0.0 | -18.5
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p = 0.318, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.438, 95% CI 2-sided [0.086 to 2.22] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.421, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 1.793, 95% CI 2-sided [0.433 to 7.426] — [estimate comment as in outcome 6, analysis 1]

10. Secondary Outcome: Change in Percent of Patients Meeting Depression Screening Criteria
Description: Screening for depression, based on Patient Health Questionnaire (PHQ-9) screen score used to quantify presence and severity of depression. Total scores range from 0 to 27, with higher score indicating more severe depression. Meeting depression screening criteria defined as the most recent PHQ-9 score < 5, indicating no or minimal depression at the time of assessment.
Time Frame: 12 months pre and post start of care coordination
Population: Patients included in analytic comparison if they had at least one PHQ9 score in both the year pre- and post-care coordination initiation.
Measure: Number; unit: percentage of patients
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 285 | 1014 | 431 | 1685
percentage of patients | 7.4 | 4.4 | 5.1 | 3.9
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p = 0.632, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.906, 95% CI 2-sided [0.606 to 1.356] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.492, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.845, 95% CI 2-sided [0.523 to 1.366] — [estimate comment as in outcome 6, analysis 1]

11. Secondary Outcome: Change in Percent of Patients Meeting A1c Control
Description: Control criteria defined as Hemoglobin A1c < or = 7%
Time Frame: 12 months pre and post start of care coordination
Population: Patients included in analytic comparison if they had a diagnosis of diabetes and had at least one available A1c results the year pre- and post-care coordination initiation.
Measure: Number; unit: percentage of patients
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 454 | 1095 | 535 | 1213
percentage of patients | 15.2 | 6.2 | 0.6 | -1.8
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p = 0.405, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.856, 95% CI 2-sided [0.594 to 1.234] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.004, Mixed Models Analysis; Odds Ratio (OR) = 0.559, 95% CI 2-sided [0.374 to 0.834]

12. Secondary Outcome: Change in Percent of Patients Meeting Aspirin or Anti-Platelet Use Recommendations
Description: Recommendation is documented aspirin use in patients unless contraindication or exception
Time Frame: 12 months pre and post start of care coordination
Population: Patients included in analytic comparison if they had vascular disease in the year pre- and post-care coordination initiation.
Measure: Number; unit: percentage of patients
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 153 | 420 | 224 | 590
percentage of patients | 2.6 | -3.1 | 3.6 | 1.2
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p = 0.071, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.151, 95% CI 2-sided [0.02 to 1.173] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.003, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Mean Difference (Net) = 0.023, 95% CI 2-sided [0.002 to 0.268] — [estimate comment as in outcome 6, analysis 1]

13. Secondary Outcome: Change in Percent of Patients Meeting Blood Pressure Control Criteria
Description: Control defined at BP < 140/90 mm Hg (SBP/DBP)
Time Frame: 12 months pre and post start of care coordination
Population: Patients included in analytic comparison if they had a diabetes and/or vascular disease diagnosis and at least one blood pressure available the year pre- and post-care coordination initiation.
Measure: Number; unit: percentage of patients
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 427 | 1067 | 541 | 1227
percentage of patients | 3.7 | -0.8 | 3.1 | 1.7
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p = 0.557, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.884, 95% CI 2-sided [0.587 to 1.333] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.069, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Mean Difference (Net) = 0.624, 95% CI 2-sided [0.376 to 1.037] — [estimate comment as in outcome 6, analysis 1]

14. Secondary Outcome: Change in Percent of Patients Meeting Statin Use Recommendations
Description: Recommendation is documented statin use in patients unless contraindication or exception
Time Frame: 12 months pre and post start of care coordination
Population: Patients included in analytic comparison if they had vascular disease diagnosis the year pre- and post-care coordination initiation.
Measure: Number; unit: percentage of patients
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 499 | 1294 | 673 | 1567
percentage of patients | 6.0 | 5.8 | 4.3 | 4.0
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p = 0.256, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.539, 95% CI 2-sided [0.185 to 1.565] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.866, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 1.117, 95% CI 2-sided [0.308 to 4.047] — [estimate comment as in outcome 6, analysis 1]

15. Secondary Outcome: Change in Percent of Patients Reporting Current Tobacco Use
Description: Current tobacco use (tobacco includes any number of cigarettes, cigars, pipes, or smokeless tobacco)
Time Frame: 12 months pre and post start of care coordination
Population: Patients included in analytic comparison if they had a diabetes and/or vascular disease diagnosis in the year pre- and post-care coordination initiation.
Measure: Number; unit: percentage of patients
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 491 | 1271 | 656 | 1561
percentage of patients | 1.8 | 0.9 | 0.2 | -0.3
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p = 0.641, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.797, 95% CI 2-sided [0.307 to 2.069] — [estimate comment as in outcome 6, analysis 1]
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.32, Mixed Models Analysis — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.569, 95% CI 2-sided [0.187 to 1.729] — [estimate comment as in outcome 6, analysis 1]

16. Secondary Outcome: Access to Care
Description: Percent of responders reporting 'Always' or 'Usually' able to get an appointment for care they need right away on survey items assessing rating of satisfaction with access to care (CG-CAHPS) -
Time Frame: 6 to 18 months after start of care coordination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 301 | 420 | 855 | 1699
Participants | 231 | 276 | 644 | 1121
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p < .001, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = 9.3, 95% CI 2-sided [5.6 to 13] — Positive values reflect higher percentage of responders in Medical/Nursing clinics as compared to Medical/Social
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.002, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = 11, 95% CI 2-sided [4.2 to 18] — Positive values reflect higher proportion of responders in Medical/Nursing clinics as compared to Medical/Social

17. Secondary Outcome: Rating of Care Coordinator
Description: The analytic outcome is defined as the percentage of patients who rated their care coordinator as a 9 or 10 on a 0-10 scale adapted from the Clinician & Group Survey (CG-CAHPS) assessment. The rating reflects patients' overall satisfaction with their care coordinator. Higher scores (9 or 10) indicate a more positive assessment of care coordination, while lower scores suggest less favorable experiences. This measure is limited to patients who recalled a recent interaction with their care coordinator.
Time Frame: 6 to 18 months after start of care coordination
Population: Patients included in analytic comparison if they responded to patient survey sent at least 6 months after care coordination initiation date , reported recent interaction with care coordinator, provided answer to relevant survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 155 | 205 | 535 | 1171
Participants | 97 | 128 | 317 | 623
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p = 0.023, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = 6.0, 95% CI 2-sided [0.86 to 11.0] — Positive values reflect higher percentage of responders in Medical/Nursing clinics as compared to Medical/Social
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.5, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = -3.7, 95% CI 2-sided [-14.0 to 7.0] — Positive values reflect higher proportion of responders in Medical/Nursing clinics as compared to Medical/Social

18. Secondary Outcome: Shared Decision Making
Description: Self-reported experience of shared decision making as measured by CollaboRATE scale - Ranges 0 to 4 higher scores represented more favorable rating of SDM
Time Frame: 6 to 18 months after start of care coordination
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 331 | 471 | 920 | 1838
score on a scale | 2.9 (0.91) | 2.7 (0.99) | 3.0 (0.89) | 2.89 (0.9)
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Mean Difference (Net) = 0.13, 95% CI 2-sided [0.06 to 0.19] — Positive values reflect higher/better scores of responders in Medical/Nursing clinics as compared to Medical/Social
Statistical Analysis 2: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p < 0.001, t-test, 2 sided — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Mean Difference (Net) = 0.19, 95% CI 2-sided [0.06 to 0.32] — Positive values reflect higher/better scores of responders in Medical/Nursing clinics as compared to Medical/Social

19. Secondary Outcome: Perceived Care Integration
Description: Self-reported experience of care integration as measured by IntegRATE scale - Ranges 0 to 3 lower scores represent more favorable rating of care integration
Time Frame: 6 to 18 months after start of care coordination
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 331 | 469 | 922 | 1832
score on a scale | 0.59 (0.54) | 0.71 (0.62) | 0.64 (0.59) | 0.75 (0.62)
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p < 0.001, t-test, 2 sided; No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.16 to -0.06] — Negative values reflect lower/better scores of responders in Medical/Nursing clinics as compared to Medical/Social
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.006, t-test, 2 sided; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.2 to -0.03] — Negative values reflect lower/better scores of responders in Medical/Nursing clinics as compared to Medical/Social

20. Secondary Outcome: Going Without Care Due to Cost
Description: Percent of patients reporting "Yes" when asked if there was any time when you needed medical care, but did not get it because you couldn't afford it in the last 12-months to cost (NHIS)
Time Frame: 6 to 18 months after start of care coordination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 326 | 455 | 914 | 1797
Participants | 23 | 58 | 81 | 203
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p = 0.059, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = -2.4, 95% CI 2-sided [-4.9 to 0.00]
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.014, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = -5.7, 95% CI 2-sided [-10.0 to -1.3] — Positive values reflect higher percentage of responders in Medical/Nursing clinics as compared to Medical/Social

21. Secondary Outcome: Out-of-pocket Medical Costs
Description: Percent of patients reporting self reporting >$500 out-of-pocket medical costs in the past 12 months (Medical expenditure panel survey)
Time Frame: 6 to 18 months after start of care coordination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 318 | 445 | 884 | 1757
Participants | 168 | 181 | 373 | 552
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p < 0.001, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = 11.0, 95% CI 2-sided [6.8 to 15.0]
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.001, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = 12.0, 95% CI 2-sided [4.7 to 20.0] — Positive values reflect higher percentage of responders in Medical/Nursing clinics as compared to Medical/Social

22. Secondary Outcome: Medication and Care Burden
Description: Self-reported medication and care burden (modified from Treatment Burden Questionnaire) - Scores range from 0 to 100 with higher scores representing more burden/worse
Time Frame: 6 to 18 months after start of care coordination
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 329 | 463 | 908 | 1792
score on a scale | 35 (31) | 41 (32) | 38 (31) | 45 (31)
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p < .001, t-test, 2 sided — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Mean Difference (Net) = -7.6, 95% CI 2-sided [-10 to -5] — Negative values reflect lower/better scores of responders in Medical/Nursing clinics as compared to Medical/Social
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.007, t-test, 2 sided; Mean Difference (Net) = -6, 95% CI 2-sided [-10 to -2] — Negative values reflect lower/better scores of responders in Medical/Nursing clinics as compared to Medical/Social

23. Secondary Outcome: Social Needs - Housing Security
Description: Percent of patients reporting "No steady place to live" when asked to describe they current living situation (modified from CMS HRSN Screening Tool)
Time Frame: 6 to 18 months after start of care coordination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 326 | 460 | 911 | 1801
Participants | 18 | 46 | 73 | 189
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p = 0.046, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = -2.5, 95% CI 2-sided [-4.8 to -0.14] — Positive values reflect higher percentage of responders in Medical/Nursing clinics as compared to Medical/Social
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.033, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = -4.5, 95% CI 2-sided [-8.4 to -0.52] — Positive values reflect higher percentage of responders in Medical/Nursing clinics as compared to Medical/Social

24. Secondary Outcome: Social Needs - Food Security
Description: Percent of patients reporting "Often", "Sometimes", or "Rarely" when asked to describe how often they or other adults in their household eat less/skip a meal because there wasn't enough money or food - (modified from CMS HRSN Screening Tool)
Time Frame: 6 to 18 months after start of care coordination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 328 | 459 | 910 | 1807
Participants | 51 | 124 | 165 | 510
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p < 0.001, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = -10.0, 95% CI 2-sided [-13.0 to -6.8] — Positive values reflect higher percentage of responders in Medical/Nursing clinics as compared to Medical/Social
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p < 0.001, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = -11.0, 95% CI 2-sided [-17.0 to -5.6] — Positive values reflect higher percentage of responders in Medical/Nursing clinics as compared to Medical/Social

25. Secondary Outcome: Social Needs - Access to Dependable Transportation
Description: Percent of patients reporting "Yes" when asked if lack of reliable transportation has kept them from participating in ADLs (modified from CMS HRSN Screening Tool)
Time Frame: 6 to 18 months after start of care coordination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 327 | 456 | 913 | 1802
Participants | 32 | 82 | 123 | 373
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p < 0.001, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = -7.2, 95% CI 2-sided [-10.0 to -4.1] — Positive values reflect higher percentage of responders in Medical/Nursing clinics as compared to Medical/Social
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.002, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = -8.2, 95% CI 2-sided [-13.0 to -3.2] — Positive values reflect higher percentage of responders in Medical/Nursing clinics as compared to Medical/Social

26. Secondary Outcome: Insurance Coverage
Description: Percent of patients reporting "No" when asked if they have any type of health care coverage (modified from CMS HRSN Screening Tool)Self-reported insurance coverage (SHADAC survey)
Time Frame: 6 to 18 months after start of care coordination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
Number analyzed (Participants) | 327 | 458 | 906 | 1798
Participants | 18 | 36 | 49 | 159
Statistical Analysis 1: Comparison: Primary Cohort: Medical/Nursing Model vs Primary Cohort: Medical/Social Model; Test type: Superiority; p = 0.002, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = -3.4, 95% CI 2-sided [-5.5 to -1.4] — Positive values reflect higher percentage of responders in Medical/Nursing clinics as compared to Medical/Social
Statistical Analysis 2: Comparison: Historical Cohort: Medical/Nursing Model vs Historical Cohort: Medical/Social Model; Test type: Superiority; p = 0.3, Chi-squared — No adjustments for multiple comparisons. Two-sided alpha of 0.05 specified a-priori; Risk Difference (RD) = -2.4, 95% CI 2-sided [-6.1 to 1.4] — Positive values reflect higher percentage of responders in Medical/Nursing clinics as compared to Medical/Social

ADVERSE EVENTS:
Description: All-cause mortality, Serious and other Adverse Events were not collected as part of this work given the observational and retrospective nature of this study. Clinics made no changes in their care practices as a result of study participation and outcomes were observed as reported in the results section. Therefore there were no patients/units considered "at-risk" for adverse event reporting.
Arm/Group | Historical Cohort: Medical/Nursing Model | Historical Cohort: Medical/Social Model | Primary Cohort: Medical/Nursing Model | Primary Cohort: Medical/Social Model
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/79/NCT04957979/Prot_SAP_002.pdf